CLINICAL TRIAL: NCT04785196
Title: A Phase Ib/II Study of APG-115 in Combination With PD-1 Inhibitor in Patients With Advanced Liposarcoma or Other Advanced Solid Tumors
Brief Title: APG-115 in Combination With PD-1 Inhibitor in Patients With Advanced Liposarcoma or Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG115XC102
Record Dates: First submitted 2021-02-24; First posted 2021-03-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Liposarcoma; Advanced Solid Tumor
Keywords: APG-115; Toripalimab; Liposarcoma; Advanced solid tumors
MeSH Terms: conditions — Liposarcoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APG-115+Toripalimab (Experimental)
  Interventions: Drug: APG-115; Drug: Toripalimab

INTERVENTIONS:
Drug: APG-115 — Dose escalation of APG-115 in combination with label dose of toripalimab, four dose levels of APG-115 will be tested: 50, 100, 150, and 200mg. APG-115 will be administrated orally every other day (QOD) for consecutive 2 weeks (ie. dosed at Day 1, 3, 5, 7, 9, 11, and 13), with one week dosing off as 3 weeks a cycle.
Drug: Toripalimab — Toripalimab is administrated following CDE approved label dose, i.e.: 240 mg intravenous infusion at Day 1 of every 3 weeks as a cycle.

SUMMARY:
Part 1 is a phase Ib standard "3 + 3" design, will be employed to determine the MTD of APG-115 by assessing the DLT of APG-115 in combination with PD-1 inhibitor(toripalimab) in advanced solid tumors.

Part 2 is a Simon two-stage phase II study design. At RP2D of APG-115 in combination with toripalimab in advanced liposarcoma, approximately 34 patients will be treated with the combination until disease progression, unacceptable toxicity, or another discontinuation criterion is met.

DETAILED DESCRIPTION:
Part 1 is the open label, dose-escalation phase Ib portion of the study to establish an MTD/RP2D of APG-115 in combination with toripalimab. Dose levels/schedule of APG115 will be tested: 50mg, 100mg, 150mg, and 200mg, QOD with 2 weeks on 1 week off as a cycle of 21 days (3 weeks), toripalimab will administrated with label dose.

Part 2 is the phase II portion of the study to evaluate the clinical efficacy and safety of the RP2D of APG-115 in combination with label dose of toripalimab in patients with advanced liposarcoma. In this part, Simon's two-stage design (Simon R (1989). Controlled Clinical Trials 10: 1-10.) will be used. The null hypothesis that the true response rate of combination is 30% or lower will be tested against a one-sided alternative. In the first stage, 19 patients will be accrued. If there are 3 or fewer responses in these patients, the study will be stopped. Otherwise, 15 additional patients will be accrued for a total of 34. The null hypothesis will be rejected if 7 or more responses are observed in 34 patients. This design yields a type I error rate of 0.05 and power of 90%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients age ≥18 years on day of signing the informed consent;
2. ECOG PS 0-1;
3. Phase Ib: Histologically confirmed, advanced liposarcoma or advanced solid tumor patients who failed standard of care therapy; Phase II: Histologically confirmed, advanced liposarcoma with TP53 wide-type and MDM2 Amplification;
4. The expected survival period is more than 12 weeks;
5. Measurable disease on CT or MRI by RECIST 1.1.
6. Adequate bone marrow and organ function as indicated by: the following laboratory values without continuous supportive treatment (such as blood transfusion, coagulation factors and/or platelet infusion, red/white blood cell growth factor administration, or albumin infusion)

   1. ANC≥1.5 x 10^9/ L;
   2. PLT≥100 x 10^9/ L;
   3. Hgb≥90 g/L;
   4. Alb≥30 g/L;
   5. AST and AST ≤3 * ULN (for hepatic metastases, ALT and AST≤5*ULN);
   6. Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance (CCr) ≥ 50ml / min.

Exclusion Criteria:

1. Patients who have previously been treated with MDM2-p53 inhibitor;
2. Known hypersensitivity reaction to PD-(L)1 inhibitors, or any prior ≥ Grade 3 irAE;
3. Prior treatment consisted of any kinds of immunotherapies, like PD-(L)1 inhibitors, anti-PD-L2 antibodies, CTLA-4, OX-40 et.al( for phase II);
4. Has known active central nervous (CNS) metastases and/or carcinomatous meningitis;
5. Has any active or history of autoimmune disease;
6. Active infection or unexplained fever > 38.5 ° C two weeks before first dose;
7. Patients with any severe and/or uncontrolled diseases, including: hypertension and uncontrollable levels of normal anti-hypertensive medication; clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction, unstable or severe angina, or coronary artery bypass surgery, congestive heart failure (New York Heart Association (NYHA) ) > 2);active or uncontrolled serious infection (≥CTCAE 5.0 Level 2 infection);objective evidence of previous or current history of pulmonary disease; moderate to severe hepatic impairment (Child-Pugh score ≥ 10 points); moderate to severe renal impairment or psychiatric illness/social circumstances that may affect study compliance;
8. Poorly controlled arrhythmia (including QTc interval ≥450 ms for males and ≥470 ms for females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (Phase I) | 21 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 3 weeks of study treatment. These will be assessed via CTCAE version 5.0.
Recommended Phase II Dose | 21 days
  Phase I is aimed to generate data to select the recommended Phase II dose.
Overall Response Rate (Phase II) | up to 12 months
  Phase II is to assess overall response rate of APG-115 in combination with toripalimab defined as the percentage of subjects with a best overall confirmed CR or a PR at any time as per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, PhD, Principal Investigator — Shanghai East Hospital
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - Shanghai East Hospital (East Hospital affiliated to Tongji University), Shanghai